CLINICAL TRIAL: NCT03627377
Title: Multi-component Intervention for Diabetes in Adults With Serious Mental Illness (MIDAS)
Brief Title: Multi-component Intervention for Diabetes in Adults With Serious Mental Illness
Acronym: MIDAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Dilip V. Jeste, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: MH15127
Record Dates: First submitted 2018-07-05; First posted 2018-08-13 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia; Obesity; Diabetes; Lifestyle Risk Reduction; Serious Mental Illness
Keywords: Schizophrenia; Serious mental illness; Obesity; Diabetes; Lifestyle Risk Reduction
MeSH Terms: conditions — Schizophrenia; Obesity; Diabetes Mellitus; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: The investigators will employ a modified cluster-randomized stepped wedge and adaptive trial design involving 210 residents with SMI and 120 staff members from 12 RCFs. The RCFs will be divided randomly into four cohorts of three RCFs each. Each cohort will be tested over a 15-month period that includes three phases: a three-month initial control phase (no intervention, from baseline month 0 to end of month 3), a six-month intervention phase (months 4 through 9), and a six-month follow-up phase (no intervention, months 10 through 15). All the study participants will be assessed quarterly during the 15-month period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Phase (No Intervention): 3-month initial control phase (no intervention, month 1-3)
- Intervention Phase (Experimental): 6-month intervention phase - MIDAS Intervention Delivered. Followed by 6-month follow-up phase (no intervention, months 10-15).
  Interventions: Behavioral: Multi-component Intervention for Diabetes in Adults with Serious Mental Illness

INTERVENTIONS:
Behavioral: Multi-component Intervention for Diabetes in Adults with Serious Mental Illness — Main components of MIDAS include: (1) Education about diabetes and lifestyle, (2) Dietary intervention at the facility and resident level, (3) Increased physical activity, and (4) Smoking cessation / reduction.
  Arms: Intervention Phase

SUMMARY:
Persons with schizophrenia and other serious mental illnesses have a high risk for type 2 diabetes and an increased risk of premature mortality compared to the general population. The goals of the proposed study are to implement a multimodal lifestyle intervention to reduce that risk in these individuals living in residential care facilities, a common housing modality for people with serious mental illnesses. If successful, this intervention will lead to reduction in excess medical comorbidity and mortality in persons with serious mental illnesses.

DETAILED DESCRIPTION:
Serious mental illnesses (SMI), including schizophrenia, bipolar disorder, and schizoaffective disorder, are associated with increased medical comorbidity and premature mortality from diabetes and cardiovascular disease. Unhealthy lifestyles, including energy-dense (obesogenic) diet, sedentary behavior, and cigarette smoking are important risk factors for diabetes and accelerated biological aging. All of these risk factors are potentially modifiable. There is considerable literature documenting the effectiveness of strategies to prevent and manage diabetes in the general population; yet, these interventions are rarely offered to people with SMI. Residential Care Facilities (RCFs), called Board-and-Care Homes in California, are a common housing modality for patients with SMI; they provide a venue that can maximize efficiency and sustainability of a lifestyle intervention. The goals of the proposed four-year study are to tailor a multi-component intervention to this high-risk group. The study will be a hybrid effectiveness-implementation (Hybrid Type 1) trial of a Multi-component Intervention for Diabetes risk reduction in Adults with SMI (MIDAS) in licensed RCFs in San Diego county. As a Hybrid Type 1 study, the primary emphasis will be on determining the effectiveness of the intervention to achieve desired health outcomes while also systematically collecting data on its implementation within RCFs that will inform implementation strategy refinement. Main components of MIDAS include: (1) Education about diabetes and lifestyle, (2) Dietary intervention at the facility and resident level, (3) Increased physical activity, and (4) Smoking cessation / reduction. The investigators will employ a modified cluster-randomized stepped wedge and adaptive trial design involving 210 residents with SMI and 120 staff members from 12 RCFs. The RCFs will be divided randomly into four cohorts of three RCFs each. Each cohort will be tested over a 15-month period that includes three phases: a three-month initial control phase (no intervention, from baseline month 0 to end of month 3), a six-month intervention phase (months 4 through 9), and a six-month follow-up phase (no intervention, months 10 through 15). All the study participants will be assessed quarterly during the 15-month period. Our investigators will train RCF staff (especially the Activity Director and cook) to increase physical activity and reduce smoking, and to implement healthful dietary modifications among the residents, using evidence-based interventions. During the intervention phase, the RCF Activity Director will conduct twice-weekly manualized group sessions on education about diabetes, nutrition, exercise, and smoking cessation/reduction, to deliver a multi-component group intervention. We will also explore if there are improvements in blood-based research biomarkers of insulin resistance and inflammation in the RCF residents with SMI. This project is responsive to RFA-MH-17-608, and related to NIMH Strategic Objective #3.3B: testing interventions for effectiveness in community practice settings. If successful, MIDAS will be sustained and disseminated, and would lead to reduction in excess medical comorbidity and mortality associated with SMI.

ELIGIBILITY:
Participants: A total of 12 RCFs (30 to 45 beds each), 210 resident participants, and 120 staff members (1 manager, 2 activity directors, 1 cook, and 6 other staff members per facility) will be enrolled.

Inclusion and Exclusion Criteria:

Residential Care Facilities (RCFs):

Inclusion Criteria:

1. Licensed by California Division of Social Services' Community Care Licensing
2. Serves only individuals with SMI
3. Has >15 residents currently living in the facility
4. Willing to participate

Staff Participants:

Inclusion Criteria:

1. Age >21 years
2. Fluent in English
3. Written informed consent to participate

Exclusion Criteria:

(1) Plans to leave the RCF during the next year.

Resident Participants:

Inclusion Criteria:

1. Age 18 - 65 years
2. Chart diagnosis of an SMI, mainly schizophrenia, schizoaffective disorder, or bipolar disorder
3. Current treatment with antipsychotics
4. Fluent in English
5. Written informed consent to participate in this study

Exclusion Criteria:

1. Chart diagnosis of dementia or intellectual disability disorder
2. Active substance abuse (non-tobacco)
3. Medical problems that interfere with ability to complete assessments and intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2018-12-28 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI in kg/m^2) | Baseline to 9 months and sustained at 15 months
  Change in Body Mass Index
Waist Circumference | Baseline to 9 months and sustained at 15 months
  Change in Waist Circumference
Fasting Glucose | Baseline to 9 months and sustained at 15 months
  Change in Fasting Glucose
Hemoglobin A1c or HbA1c | Baseline to 9 months and sustained at 15 months
  Change in Hemoglobin A1c or HbA1c

SECONDARY OUTCOMES:
Diet/Nutrition - Plasma Carotenoid Levels | Baseline to 9 months and sustained at 15 months
  Plasma Carotenoid levels reflect changing dietary vegetable and fruit intake.Nutrition Data Systems for REsearch (NDS-R) Protocol
Diet/Nutrition - Serum Lipid Levels | Baseline to 9 months and sustained at 15 months
  Plasma Carotenoid levels reflect changing dietary vegetable and fruit intake.
Objective Measure of Physical Activity | Baseline to 9 months and sustained at 15 months
  For 7 days during each assessment period, participants will wear the GT3X+ Actigraph, which measures movement and intensity of activity, and has good validation with VO2max. It provides estimates of activity by seconds, that can be categorized into minutes spent in sedentary, light, moderate, and vigorous activity using calibration thresholds.
Smoking - Expired Breath Carbon Monoxide (CO) Levels | Baseline to 9 months and sustained at 15 months
  Change in Smoking - Objective Measure of Cigarette Use: Expired Breath Carbon Monoxide (CO) level (parts per million) is measured with a handheld device. CO monitoring is used primarily as a check on recent smoking, though it has also been used to indicate reductions in smoking.
Smoking - Change in Smoking through Recall | Baseline to 9 months and sustained at 15 months
  Change in Smoking - Quantity and frequency of cigarette use for the prior week using a timeline followback procedure. Smoking reduction calculated by % change in average cigarettes/day across assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego Division of Geriatric Psychiatry, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No